CLINICAL TRIAL: NCT07386925
Title: Clinical and Radiographic Evaluation of Pelargonium Graveolens Essential Oil as a Pulpotomy Agent in Primary Teeth
Brief Title: Pelargonium Graveolens Essential Oil as a Pulpotomy Agent in Primary Teeth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shaimaa Shaban Mohamed El-desouky, assistant professor of pediatric dentistry, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: # R-PED-12-25-3237
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Pulpitis - Reversible; Pulpotomies on Primary Molars
Keywords: Pelargonium graveolens; pulpotomy; MTA
MeSH Terms: interventions — Pulpotomy; Radiation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: zinc oxide-geranium (Pelargonium graveolens) essential oil paste (Experimental): 30 primary molars will be treated with geranium (Pelargonium graveolens) essential oil freshly mixed with zinc oxide powder till it reaches a suitable consistency (1:1 ratio by volume) to cover pulp stumps
  Interventions: Procedure: pulpotomy; Procedure: Radiation
- group 2: MTA (Active Comparator): 30 primary molars will be treated with MTA to cover pulp stumps
  Interventions: Procedure: pulpotomy; Procedure: Radiation

INTERVENTIONS:
Procedure: pulpotomy — Teeth will be anesthetized then Rubber dam and high suction will be used in pulpotomy procedure. Cavity outline will be performed by sterile #330 high speed bur using water spray. Caries will be removed by large spoon excavator. When pulpal exposure occurred, the roof of pulp chamber will be removed by low speed round bur. Haemostasis will be obtained by applying pressure with a moist cotton pellet with saline. Then the test materials will be applied. after that, pulp stumps of all molars in each group will be dressed using Intermediate restorative material, then the tooth will be restored with a preformed stainless steel crown
Procedure: Radiation — Radiographic evaluation will be performed immediately after teeth restoration (baseline radiograph), then after three, six, and twelve months for the furcation radiolucency area and bone radiodensity. A photo-simulated phosphorus plate sensor was used to take direct standardized digital radiographs. The parallel periapical technique was obtained by Rinn, which is attached to the X-ray tube with its arm fastened to the film holder that contained a coated PSP (photo-stimulated phosphorus plate). To ensure standardization during radiographic film retakes, condensation rubber base impression material will be positioned on the outside of the film holder, and the child is told to bite on it while the material is set. The sensor wil exposed to an X-ray machine (Planmeca ProX, Helsinki, Finland) with a central ray perpendicular to the sensor at 70 kVp, 6 mA, and 0.8 s. Radio-densitometric and radiometric analysis of the radiographs will be performed by RadiAnt software.

SUMMARY:
The success of pulpotomy in primary teeth is critical for preserving function and arch integrity in children and depends largely on the biological properties of the medicament used. Given the limitations of mineral trioxide aggregate, Pelargonium graveolens essential oil has emerged as a potential alternative; however, its clinical performance as a pulpotomy agent remains insufficiently investigated.

DETAILED DESCRIPTION:
The use of medicinal plants and herbal extracts in modern dentistry is steadily increasing, primarily due to their antimicrobial properties and high biocompatibility. Pelargonium graveolens (rose geranium), native to South Africa, produces an essential oil rich in geraniol, citronellol, and linalool[18]. Geraniol, present in rose geranium oil, is recognized for its antioxidant, anti-inflammatory, antimicrobial, and anticancer effects. The oil's main constituents, beta-citronellol and geraniol, contribute to its antifungal and wound-healing properties, making it a promising agent for treating denture-induced stomatitis

ELIGIBILITY:
Inclusion Criteria:

* Restorable primary molars with deep carious lesions.
* Absence of gingival swelling or sinus tract.
* Absence of spontaneous pain
* Absence of pain on percussion.
* Absence of discontinuity of lamina dura
* Absence of internal root resorption.
* Absence of external root resorption.
* Absence of inter-radicular or periapical bone destruction (radiolucency).

Exclusion Criteria:

* presence of spontaneous pain
* presence of gingival swelling or sinus tract
* presence of internal or external root resorption
* pain on percussion.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
absence of pain | up to 9 months
  Measuring Method: Verbal Question to Patient /Parents Measuring Unite: score 0 for absence of pain and score 1 for presence of pain
absence of fistula | up to 9 months
  Measuring Method: Visual examination by operator Measuring Unit: score 0 for absence of swelling and score 1 for presence of swelling
Tenderness to percussion | up to 9 months
  Measuring Method: Percussion test Measuring Unite: Binary (+/-)
Furcation radiolucency | 3 months
  Measuring Method: periapical x-ray for assessment of radio-density of bone at the furcation area, Measuring Unit: mean value of gray level (which measures density scale between 0 to 256, with zero being the lowest value and 256 the highest dense value)
furcation radiolucency | 6 months
  Measuring Method: periapical x-ray for assessment of radio-density of bone at the furcation area, Measuring Unit: mean value of gray level (which measures density scale between 0 to 256, with zero being the lowest value and 256 the highest dense value)
furcation radiolucency | 9 months
  Description: Measuring Method: periapical x-ray for assessment of radio-density of bone at the furcation area, Measuring Unit: mean value of gray level (which measures density scale between 0 to 256, with zero being the lowest value and 256 the highest dense value)

CONTACTS AND LOCATIONS:
Overall Officials: shimaa Hadwa, Principal Investigator — shimaa.hadwa@dent.tanta.edu.eg
Locations (1):
- faculty of dentistry, Tanta university, Tanta, Egypt

REFERENCES:
- [Background] Holan, G., E. Eidelman, and A.B. Fuks, Long-term evaluation of pulpotomy in primary molars using mineral trioxide aggregate or formocresol. Pediatric dentistry, 2005. 27(2): p. 129-136
- [Background] Subramanyam, D. and S. Somasundaram, Clinical and radiographic outcome of herbal medicine versus standard pulpotomy medicaments in primary molars: a systematic review. J Clin Diagn Res, 2017. 11(10): p. ZE12-ZE16.